CLINICAL TRIAL: NCT07316023
Title: Efficacy of Antimicrobial Photodynamic Therapy Using Polymeric Nanoparticles Loaded With Indocyanine Green in Management of Periodontitis.(A Randomized Controlled Clinical Trial Study With Microbiological Analysis )
Brief Title: Antimicrobial Photodynamic Therapy With ICG-Loaded Nanoparticles for Periodontitis Management
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nada Mahmoud Soliman (Other)
Responsible Party: Sponsor-Investigator, Nada Mahmoud Soliman, master Candidate at oral medicine and periodontology department faculty of dentistry ainshams university, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Polymeric Nanoparticles /ICG
Record Dates: First submitted 2025-11-16; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Stage III Periodontitis
Keywords: periodontits/ stage III / NSPT/PDT/Nano particles/ ICG
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated using computer-generated randomization (www.Randomizer.org
  ) into three groups of nine each. Group I will receive non-surgical periodontal therapy (NSPT) combined with ICG-loaded polymeric nanoparticles and antimicrobial photodynamic therapy (aPDT). Group II (positive control) will receive NSPT with ICG gel and aPDT, while Group III (negative control) will receive NSPT alone. After full-mouth debridement and baseline GCF and clinical data collection, the photosensitizer will be applied for 10 minutes, followed by diode laser irradiation (940 nm, 0.5 W, continuous mode, 30 seconds per site using a 0.3 nm E3 tip in contact mode). Excess gel will be removed after activation, and aPDT will be performed once. All patients will receive oral hygiene instructions, and clinical and GCF evaluations will be conducted at baseline, immediately post-treatment, 1 week, 1 month, 3 months, and 6 months.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nano Group (Experimental): This group will include 9 patients diagnosed with generalized stage III periodontitis and will be treated with non-surgical periodontal treatment + ICG-loaded polymeric nanoparticles + antimicrobial photodynamic therapy (aPDT).
  Interventions: Drug: Non- surgical periodontal therapy followed by photodynamic therapy with ICG-loaded nanoparticles
- Macro Group( positive control) (Active Comparator): Group (II): Positive Control This group will include 9 patients diagnosed with generalized stage III periodontitis and will be treated with non-surgical periodontal treatment + ICG gel application alone + antimicrobial photodynamic therapy.
  Interventions: Drug: Non- surgical periodontal therapy followed by photodynamic therapy with ICG-loaded macroparticles
- Negative Control (Other): Group (III): Negative Control This group will include 9 patients diagnosed with stage III periodontitis and will be treated with non-surgical periodontal therapy only.
  Interventions: Other: Non- surgical periodontal therapy only

INTERVENTIONS:
Drug: Non- surgical periodontal therapy followed by photodynamic therapy with ICG-loaded nanoparticles — Supragingival scaling and subgingival debridement followed by placement of ICG-loaded nanoparticles activated by diode laser for antibacterial photodynamic therapy to effectively target and eliminate pathogenic bacteria.
  Arms: Nano Group
Drug: Non- surgical periodontal therapy followed by photodynamic therapy with ICG-loaded macroparticles — supragingival scaling and subgingival debridement followed by ICG-loaded macroparticles activated by diode laser for antibacterial photodynamic therapy to effectively target and eliminate pathogenic bacteria.
  Arms: Macro Group( positive control)
Other: Non- surgical periodontal therapy only — supragingival scaling and subgingival debridement only
  Arms: Negative Control

SUMMARY:
To better understand and treat your gum disease, dentists now use a system that stages its severity and grades its speed, rather than using old labels. The recommended first step is almost always a deep cleaning, which is very effective. However, because some bacteria can hide from cleanings and antibiotics, researchers are exploring a promising light-based treatment. This method uses a safe, light-activated dye and a gentle laser to target and kill bacteria without leading to resistance. To make this treatment even stronger, scientists are testing a way to package the dye inside tiny, biodegradable "containers" that deliver it directly to the germs. The goal of this research is to see if this advanced delivery method works better than the dye alone, hoping to provide a more powerful, non-surgical option to fight gum disease and protect your teeth."

DETAILED DESCRIPTION:
This randomized controlled clinical trial included twenty-seven patients diagnosed with generalized stage III periodontitis, who were randomly allocated into three groups using a computer-generated randomization sequence (www.randomizer.org

). Group I (test group) received non-surgical periodontal therapy followed by the application of indocyanine green (ICG)-loaded polymeric nanoparticles and antimicrobial photodynamic therapy (aPDT). Group II (positive control) received non-surgical periodontal therapy with ICG gel application alone and aPDT, whereas Group III (negative control) received non-surgical periodontal therapy only. Following full-mouth supra- and subgingival debridement, baseline clinical measurements and gingival crevicular fluid (GCF) samples were obtained. In Groups I and II, after achieving site dryness, the photosensitizer was applied for 10 minutes, rinsed, and activated using a 940 nm diode laser (0.5 W, continuous mode, non-initiated E3 tip, contact mode, 30 seconds per site, six sites per tooth). Standardized oral hygiene instructions were provided to all participants. Clinical and microbiological evaluations were performed at baseline, 3 months, and 6 months post-treatment. Clinical parameters including plaque index, gingival index, probing depth, and clinical attachment level were recorded using a UNC-15 probe. For microbiological analysis, GCF samples from the most affected sites were collected at baseline, immediately post-treatment, 1 week, and 1 month, and analyzed by polymerase chain reaction (PCR) to quantify Porphyromonas gingivalis. Samples contaminated with blood or saliva were excluded, and uncontaminated samples were transported in reduced transport fluid (RTF) and cultured under anaerobic conditions for bacterial quantification.

The obtained results will be collected, tabulated, and subjected to appropriate statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* 1- Both genders aged between 36-50 years (Wadhwa et al., 2021) 2- Generalized stage III grade B periodontitis (Papapanou et al., 2018). Posterior teeth, stage III with PD>6 mm and CAL ≥5 mm 3- Patients ready to comply with oral hygiene measures. 4- Patients free from any systemic disease that may affect the treatment (Glick et al., 2008)

Exclusion Criteria:

* Exclusion criteria:

  1. Smokers
  2. Pregnant females.
  3. Drug abusers.
  4. Patients taking antibiotics or performed any periodontal treatment in the previous 6 months.

Justification for Exclusions:

To reduce any confounding factors and bias that may affect the results of this study.

Ages: 36 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Plaque Index (unit:score) | from the enrollment to the end of treatment at 6 months the clinical parameters are first measured at baseline through stent for standaridization and then measured again after 3 months and 6 months repectively .
  Clinical parameters including plaque index, gingival index, probing pocket depth (PPD), and clinical attachment level (CAL) will be recorded at baseline, 3, and 6 months using a UNC-15 probe by a calibrated examiner. The plaque and gingival indices (Löe and Silness, 1963) assess oral hygiene and inflammation. The following clinical parameters will be taken using the UNC15 Probe at baseline, 3 months, and 6 months postoperative.
  - Plaque index: - (Loe and Silness, 1963) 0 = no plaque.
  1. = plaque recognized only by running a probe across the marginal surface of implant restoration.
  2. = plaque visible to the naked eye.
  3. = abundance of soft matter.
The Gingival index (unit=score ) | from the enrollment to the end of treatment at 6 months the clinical parameters are first measured at baseline through stent for standaridization and then measured again after 3 months and 6 months repectively .
  The following clinical parameters will be taken using UNC15 Probe at baseline, 3 months and 6 months postoperative.
  - Gingival index: -(Loe and Silness ,1963) 0 = Normal gingiva
  1. = Mild inflammation - slight edema. No bleeding on probing
  2. = Moderate inflammation -redness, edema and glazing. Bleeding on probing.
  3. = Severe inflammation - marked redness and edema. Ulceration. Tendency to spontaneous bleeding
Probing depth (PD) (Unit=mm) | from the enrollment to the end of treatment at 6 months the clinical parameters are first measured at baseline through stent for standaridization and then measured again after 3 months and 6 months repectively .
  Will be measured from the gingival margin to the depth of the pocket at four points (mesio-facial, mid-facial, disto-facial and mid-lingual) to the nearest millimeter using UNC-15 periodontal probe The average of the three facial points will be recorded as the facial probing depth (FPD), while the mid-lingual point will be recorded as the lingual probing depth.
Clinical Attachment Loss (CAL) (Unit=mm) | from the enrollment to the end of treatment at 6 months the clinical parameters are first measured at baseline through stent for standaridization and then measured again after 3 months and 6 months repectively .
  - Clinical attachment level (CAL): (Ramfjord et al., 1975). Will be measured from the CEJ to the depth of the periodontal pocket.

SECONDARY OUTCOMES:
Microbial evaluation to detect bactericidal effect on Porhyromonas gingivalis. | from enrollment to the end of treatment at 6 months GCF samples will be collected from the deepest, most affected sites at baseline line , immediate postlaser treatment and after one month respectively
  Microbiological analysis will assess P. gingivalis levels in gingival crevicular fluid (GCF) using PCR at baseline, immediately post-treatment, one week, and one month. GCF samples will be collected from the most affected site using sterile paper strips, avoiding blood or saliva contamination, and stored in reduced transport fluid. Samples will be cultured and analyzed by PCR for P. gingivalis quantification. Results will compare microbial reduction among groups to evaluate the antimicrobial efficacy of nano- and macro-formulated photosensitizer gels versus conventional debridement.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry , Ainshams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No